CLINICAL TRIAL: NCT02799849
Title: Is There a Change in the Total Metabolism Over 24 Hours for Narcoleptic Children That Could Explain Their Tendency to Obesity?
Brief Title: Metabolism Characteristics in the Children With Narcolepsy
Acronym: Narcolepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-759
Record Dates: First submitted 2016-05-03; First posted 2016-06-15 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Narcolepsy
Keywords: narcolepsy; metabolism
MeSH Terms: conditions — Narcolepsy | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narcoleptic patients (Other)
  Interventions: Other: Sleep and metabolism assessment
- hypersomnic patients (Other)
  Interventions: Other: Sleep and metabolism assessment

INTERVENTIONS:
Other: Sleep and metabolism assessment

SUMMARY:
A significant weight gain and obesity are observed for most patients with narcolepsy, mainly at the beginning of the disease and narcolepsy in young children. There is no specific study on the population and the consequences of overweight in the lives of these long-term patients. Narcoleptic patients gain weight significantly at the onset of their illness. It is also known that weight gain is not related to the treatment of narcolepsy. The etiology of obesity in narcoleptic patients is not established. Several assumptions were made (physical activity, leptin diet, metabolism). The reason and the pathophysiology of overweight and obesity in this population therefore remain unclear.

In this study, potential change in the total metabolism (24h) for narcoleptic children that could explain their tendency to obesity will be assessed ?

ELIGIBILITY:
Inclusion Criteria:

NARCOLEPTIC PATIENTS

* Girl or boy age> 6 years <18 years;
* Narcoleptic: defined by the ICSD diagnostic criteria 2 (International Classification of Sleep Disorders)
* Beginning of the troubles there more than 6 months
* Parental consent and agreement of the child.

HYPERSOMNIC PATIENTS

* Girl or boy age> 6 years <18 years;
* Hypersomnic : defined by the ICSD diagnostic criteria 2 (International Classification of Sleep Disorders)
* Beginning of the troubles there more than 6 months
* Parental consent and agreement of the child.

Exclusion Criteria:

NARCOLEPTIC PATIENTS

* Secondary Narcolepsy;
* Narcolepsy already treated with psychostimulant or anticataplectic;
* Restless legs;
* Sleep apnea syndrome;
* Obesity known outside narcolepsy cause;
* Absence of parental consent.

HYPERSOMNIC PATIENTS

* symptomatic or secondary hypersomnia;
* Hypersomnia already treated psychostimulant or anticataplectic; Restless legs;
* Sleep apnea syndrome;
* Pathology neurological, psychiatric, endocrine or concurrent;
* Lack of parental consent

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12-20 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Determination of the metabolism at home | 15 days
  Total energy expenditure in kilocalories per minute, including basal metabolic rate (MET) metabolism related to the activity (EEA), and physical activity (PA) measured by accelerometer (Actical) evaluated at home (15 days including scholar and non-scholar days).

SECONDARY OUTCOMES:
Determination of the metabolism at hospital | 18 days
  Total energy expenditure in kilocalories per minute, including basal metabolic rate (MET) metabolism related to the activity (EEA), and physical activity (PA) measured by accelerometer (Actical) evaluated at hospital over 24 hours.
Basal energy expenditure | 18 days
  The basal metabolism (MET) measured by accelerometer (Actical, BodyMedia SW Actiheart) will be compared to the values of energy expenditure (kcal) measured by indirect calorimetry fasting.
Energy expenditure and diet-induced thermogenesis | 18 days
  Energy expenditure (kcal) measured by indirect calorimetry after lunch (with counting calories ingested).
Sympathetic activity | 18 days
  Estimated from IBI (Interbeat Interval) measured by Actiheart.
Food intake | 18 days
  Caloric intake evaluation (kcal per day) during hospitalization (food intake recording) and at home during three days ( two days during the week and one day during the week-end) evaluated by questionnary.
Fasting peptide YY | 18 days
Body weight | 18 days
  bodyweight (kg)
Body height | 18 days
  Body height (cm)
Waist and hips circumference | 18 days
  Waist and hips circumference (cm)
Measurement of neck | 18 days
  Measurement of neck (cm)
Anthropometric measurements | 18 days
  Measurement of BMI Z-score
Appetite | 18 days
  appetite evaluation by visual analog scale before each meal
Hunger | 18 days
  hunger evaluation by visual analog scale before each meal
Fasting IL6-8 levels | 18 days
Fasting adiponectin | 18 days
Fasting resistin | 18 days
Fasting MCP1 | 18 days
Fasting PostPrandial | 18 days
Fasting GLP1 (glucagon-like peptide-1) | 18 days
Fasting Hba1C | 18 days
Body mass index z score | 18 days
sleep duration | 18 days

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Exploration et pathologie du sommeil, Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No